CLINICAL TRIAL: NCT06991829
Title: Clinical Study on the Safety and Efficacy of Immunophenotyped Pancreatic Endocrine Organoid Bank in Treating Patients With T3c Diabetes
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Newislet Therapeutics Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-10
Record Dates: First submitted 2025-04-15; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: type 3c diabetes mellitus; pancreatic endocrine organoids; Islet Transplantation; HLA-immunotyped
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A single-arm clinical trial is designed to evaluate whether transplantation of HLA-matched pancreatic endocrine organoids can effectively lower blood glucose levels in patients with diabetes following pancreatectomy. The trial employs Simon's Two-Stage Optimal Design to determine sample size, with parameters: P0 = 0.10 (null hypothesis), P1 = 0.30 (alternative hypothesis), α = 0.05, and β = 0.20. Given the lack of definitive treatments and the first-in-human nature of this intervention, 10 patients will be enrolled in the first stage. If ≥2 achieve treatment success, the trial proceeds to stage two; otherwise, it stops. In stage two, 19 more patients will be enrolled (total n=29). If ≥6 patients achieve treatment success, the therapy is considered effective; if <6, it is considered ineffective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLA-matched pancreatic endocrine organoids transplantation (Experimental): Islet cells are isolated from resected pancreatic tissue obtained from patients undergoing surgery, followed by ex vivo expansion and culture. Subsequent procedures include HLA typing, functional assessment of organoid-like structures, and biobanking. After matching for HLA, the cells are administered into patients with type 3c diabetes mellitus (T3cDM) via ultrasound-guided percutaneous transhepatic portal vein catheterization. A 52-week follow-up is conducted to evaluate the safety of the cell therapy and its clinical efficacy in glycemic control.
  Interventions: Procedure: HLA-matched pancreatic endocrine organoids transplantation

INTERVENTIONS:
Procedure: HLA-matched pancreatic endocrine organoids transplantation — Islet cells are isolated from resected pancreatic tissue obtained from patients undergoing surgery, followed by ex vivo expansion and culture. Subsequent procedures include HLA typing, functional assessment of organoid-like structures, and biobanking. After matching for HLA, the cells are administered into patients with type 3c diabetes mellitus (T3cDM) via ultrasound-guided percutaneous transhepatic portal vein catheterization. A 52-week follow-up is conducted to evaluate the safety of the cell therapy and its clinical efficacy in glycemic control.

SUMMARY:
Islet cells are isolated from resected pancreatic tissue obtained from patients undergoing surgery, followed by ex vivo expansion and culture. Subsequent procedures include HLA typing, functional assessment of organoid-like structures, and biobanking. After matching for HLA, the cells are administered into patients with type 3c diabetes mellitus (T3cDM) via ultrasound-guided percutaneous transhepatic portal vein catheterization. A 52-week follow-up is conducted to evaluate the safety of the cell therapy and its clinical efficacy in glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤70 years at the time of informed consent, regardless of sex; History of total pancreatectomy with baseline C-peptide levels below the lower limit of normal;
2. Post-pancreatectomy hyperglycemia consistent with diagnostic criteria for T3cDM;
3. Stimulated C-peptide level < 0.3 ng/mL at 120 minutes following a mixed meal;
4. HbA1c≥7.5% or TIR < 70% despite intensified insulin therapy;
5. Male participants who are sexually active and not surgically sterilized or whose partners are of childbearing potential must agree to use effective contraception and refrain from sperm donation throughout the study and for at least 6 months thereafter; female participants of childbearing potential must agree to use effective contraception for the duration of the study and for at least 6 months thereafter.
6. Voluntary written informed consent and willingness to comply with the study protocol and visit schedule.

Exclusion Criteria:

1. Known hemoglobinopathies or moderate-to-severe anemia interfering with HbA1c interpretation;
2. Positive HBsAg or HBcAb with HBV DNA ≥10⁴ copies/mL or ≥2000 IU/mL; Patients with positive HBsAg and HBV DNA <2000 IU/mL must be on antiviral therapy throughout the study. Patients with positive HBcAb and HBV DNA <2000 IU/mL must undergo regular HBV DNA monitoring;
3. Positive HCV antibody with HCV RNA≥10³IU/mL;
4. Positive HIV antibody testing;
5. Active syphilis infection (those with resolved infection may be included);
6. Existence or suspicion of other uncontrollable or untreatable fungal, bacterial, viral or other infections;
7. Uncontrolled hypertension (SBP >160 mmHg and/or DBP >100 mmHg despite stable antihypertensive treatment for ≥4 weeks);
8. History of coagulopathy or long-term anticoagulation therapy (e.g., warfarin) or INR >1.5 (low-dose aspirin permitted);
9. Impaired liver function: AST or ALT >3× ULN Total bilirubin >2× ULN;
10. Impaired renal function with Creatinine clearance <45 mL/min (Cockcroft-Gault formula);
11. History of end-stage heart or lung disease, or cirrhosis;
12. Presence or history of any type of cancer, excluding papillary thyroid cancer cured for more than 1 year;
13. Severe mental/psychological disorders, or severe cognitive impairment
14. Pregnant or lactating women;
15. Other situations or abnormal findings judged by the investigator as unsuitable for participating in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04-03 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with ≥50% Reduction in Daily Insulin Dose at Week 52 Post-Transplantation Compared to Baseline | From enrollment to the end of treatment at 52 weeks post-transplantation
  The percentage of participants whose daily insulin requirement is reduced by at least 50% at 52 weeks after organoid transplantation, compared to their baseline insulin dose.
Proportion of Participants with HbA1c < 7.0% at Week 52 Post-Transplantation | From enrollment to the end of treatment at 52 weeks post-transplantation
  The percentage of participants achieving HbA1c levels <7.0% at 52 weeks post-transplantation, indicating improved long-term glycemic control.
Number of Participants with No Episodes of Severe Hypoglycemia Between Weeks 12 and 52 Post-Transplantation | From Week 12 to Week 52 post-transplantation
  The number of participants who report zero episodes of severe hypoglycemia during the 12 to 52 weeks post-transplantation period.

SECONDARY OUTCOMES:
Proportion of Participants with HbA1c < 7.0% at Weeks 12, 26, and 52 Post-Transplantation | Weeks 12, 26, and 52 post-transplantation
  Percentage of participants achieving HbA1c < 7.0% at each follow-up time point to assess glycemic control over time.
Proportion of Participants with ≥50% Reduction in Daily Insulin Dose at Weeks 12, 26, and 52 Post-Transplantation | Weeks 12, 26, and 52 post-transplantation
  Percentage of participants whose insulin requirement is reduced by at least 50% at three time points post-transplantation.
Proportion of Participants Achieving Insulin Independence at Weeks 26 and 52 Post-Transplantation | Weeks 26 and 52 post-transplantation
  Percentage of participants who achieve complete insulin independence by Week 26 and Week 52.
Proportion of Participants with Stimulated C-Peptide Peak > 0.3 ng/mL Following a Mixed Meal Tolerance Test at Weeks 12, 26, and 52 | Weeks 12, 26, and 52 post-transplantation
  Percentage of participants with stimulated C-peptide > 0.3 ng/mL at Weeks 12, 26, and 52, indicating β-cell functional recovery.
Time-in-Range (TIR) at Weeks 12, 26, and 52 Post-Transplantation | Weeks 12, 26, and 52 post-transplantation
  Proportion of time during which blood glucose levels remain within target glycemic range, as measured by CGM.
Mean Amplitude of Glycemic Excursions (MAGE) at Weeks 12, 26, and 52 Post-Transplantation | Weeks 12, 26, and 52 post-transplantation
  Glycemic variability measured by the average amplitude of glucose excursions as recorded by CGM.
Cumulative Number of Hypoglycemic Episodes at Weeks 12, 26, and 52 Post-Transplantation | Weeks 12, 26, and 52 post-transplantation
  Number of documented hypoglycemic events recorded during follow-up.
Number of Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) | From enrollment to Week 52 post-transplantation.
  Safety profile assessed by the number and type of adverse events recorded over the treatment period.
Change in Quality of Life Scores from Baseline to Week 52 Post-Transplantation | From enrollment to the end of treatment at 52 weeks post-transplantation
  Difference in patient-reported quality of life scores from baseline to Week 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP) and Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Throughout the entire clinical trial period
Access Criteria: Qualified researchers who provide a methodologically sound proposal will be able to access the individual participant data (IPD) and related documents such as the study protocol and statistical analysis plan. Access will be granted through a secure data sharing platform upon request and approval by the study sponsor or a designated data access committee. All shared data will be de-identified to protect participant confidentiality.
URL: https://www.zs-hospital.sh.cn/zhuanye/channel/5429/1/205.html